CLINICAL TRIAL: NCT01072851
Title: Tools for Improving Colorectal Cancer Screening Rates: Multimedia vs Print
Brief Title: Tools for Improving Colorectal Cancer Screening Rates: Multimedia Versus Print
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Collaborators: American Cancer Society, Inc. (Other); Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0910001-E
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer screening; multimedia education; print education; culturally competent
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Patient Education as Topic; Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Multimedia educational tool (Experimental): Multimedia education tool - A culturally competent video explaining the importance of and the process of colorectal cancer screening
  Interventions: Behavioral: Multimedia Education
- Print educational tool (Experimental): Print media - A culturally competent printed brochure explaining the importance of and the process of colorectal cancer screening
  Interventions: Behavioral: Print Media
- No intervention (Active Comparator): Usual and customary waiting room process - Usual and customary office waiting period with access to standard nationally generated colorectal cancer screening informational material in the waiting room and/or exam room.
  Interventions: Behavioral: Usual and customary waiting room process

INTERVENTIONS:
Behavioral: Multimedia Education — A four minute exposure to an educational video with controlled content on the importance of colorectal cancer screening and explaining the processes and procedures.
  Other Names: colon cancer; communication; patient education
  Arms: Multimedia educational tool
Behavioral: Print Media — Exposure to a printed brochure with controlled content on the importance of colorectal cancer screening and explaining the processes and procedures.
  Other Names: colon cancer; communication; education
  Arms: Print educational tool
Behavioral: Usual and customary waiting room process — No specialized educational intervention to promote colorectal cancer screening or to explain the process
  Other Names: colon cancer; communitcation; education
  Arms: No intervention

SUMMARY:
The objective of this study is to compare the effectiveness of multimedia and print tools designed to provide patients at safety-net clinics with comprehensible information about colorectal cancer screening and motivate them to complete screening.The print and multimedia interventions were constructed with parallel content to allow valid comparison of format-related effects on knowledge and screening rates.These easy to use tools will provide under served patients at community health centers with clear and consistent messages about colorectal Cancer(CRC) and CRC screening, delivered immediately before the patients see a doctor.

Specific Aims

1. To determine if multimedia and print interventions that provide patients with information and motivational messages about CRC screening increase screening rates above usual care.
2. Determine whether showing patients a multimedia program achieves higher CRC screening rates than does a print booklet with equivalent messages.

   1. Examine if the effects of these multimedia and print interventions on CRC screening rates differ with literacy level.
   2. Examine if the effects of these multimedia and print interventions on CRC screening differ with race/ethnicity
   3. Examine if these multimedia and print interventions have differential effects on knowledge relevant to CRC screening.

DETAILED DESCRIPTION:
Despite the clear benefits of screening for early detection and prevention of colorectal cancer, as many as half of eligible adults remain unscreened. Poor and under served populations, particularly African American and Latino/Hispanic adults, are at greatest risk for noncompliance with recommended tests. Health education strategies developed to date have led to relatively minimal gains, resulting in little translation to routine clinical practice. This is especially true in more difficult, resource-strained practice settings, such as community health centers.

The interventions in the proposed study draw on communication science to optimize message design, use communication technology to optimize message delivery and include parallel content in both print and multimedia versions to allow comparison of format-related effects on both knowledge and screening rates.The multimedia and print tools are based on patient education programs that we developed with extensive attention to theory as well as community member input.

ELIGIBILITY:
Inclusion Criteria:

* 50-80 years of age,
* Registered for an appointment at one of the target clinics,
* Speaks English or Spanish.

Exclusion Criteria:

* Patient has had CRC screening in the past 12 months,
* Unable to review the study materials because of language, physical condition or literacy.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the acceptance of colorectal cancer screening by patients who view print or multimedia educational tools | 3 months post visit

SECONDARY OUTCOMES:
Role of race/ethnicity and literacy levels on the comparative effects if the intervention | At scheduled appointment
Comparative knowledge of colorectal cancer screening by patients who view the print or multi-media educational tools. | At the scheduled patient visit

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Makoul, PHD, Principal Investigator — St. Francis Hospital & Medical Center, Hartford CT
Locations (3):
- United States (3):
  - Midlakes Medical Building, Highland Park, Illinois
  - North Chicago Health Center, North Chicago, Illinois
  - Belvidere Medical Building, Waukegan, Illinois